CLINICAL TRIAL: NCT01365845
Title: Proton Therapy for Peripheral Lymph Nodes in Breast Cancer
Brief Title: Proton Therapy for Lymph Nodes in Breast Cancer
Acronym: BR01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701740; UFPTI 1016-BR01 (Other: University of Florida Project #)
Record Dates: First submitted 2011-05-19; First posted 2011-06-03 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Proton Radiation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Conventional photon plan
  Interventions: Radiation: Photon
- 2 (Experimental): 3D-Proton/Conventional plan or 3D-proton only
  Interventions: Radiation: 3D-Proton/Conventional plan or 3D-proton only

INTERVENTIONS:
Radiation: Photon — 50.4 Gy to the breast/chest wall and peripheral lymph nodes at 1.8 Gy per fraction
  Arms: 1
Radiation: 3D-Proton/Conventional plan or 3D-proton only — 50.4 Cobalt Gray Equivalent/Gray to the breast/chest wall and peripheral lymph nodes at 1.8 Cobalt Gray Equivalent/Gray per fraction
  Arms: 2

SUMMARY:
The purpose of this study is to determine if proton radiation therapy will reduce the amount of heart that is exposed to radiation, thereby decreasing the frequency and/or severity of any cardiac side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive adenocarcinoma of the breast stage I-III (TX, T0-4, N0-3) with medially located tumor and/or axillary node invasion.
* Patients must have undergone either mastectomy or breast conservation surgery.
* Patients are required to have axillary staging which can include sentinel node biopsy alone if sentinel node is negative.
* Patient must require peripheral lymph node radiation per physician discretion.

Exclusion Criteria:

* Evidence of distant metastasis (M1).
* Prior radiotherapy to the area of interest.
* Prior history of cardiovascular disease per physician discretion.
* Prior or concurrent cancer other than non-melanomatous skin cancer unless disease free for at least 5 years.
* Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis or scleroderma.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Bradley, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Overgaard M, Hansen PS, Overgaard J, Rose C, Andersson M, Bach F, Kjaer M, Gadeberg CC, Mouridsen HT, Jensen MB, Zedeler K. Postoperative radiotherapy in high-risk premenopausal women with breast cancer who receive adjuvant chemotherapy. Danish Breast Cancer Cooperative Group 82b Trial. N Engl J Med. 1997 Oct 2;337(14):949-55. doi: 10.1056/NEJM199710023371401. PMID 9395428
- [Background] Overgaard M, Jensen MB, Overgaard J, Hansen PS, Rose C, Andersson M, Kamby C, Kjaer M, Gadeberg CC, Rasmussen BB, Blichert-Toft M, Mouridsen HT. Postoperative radiotherapy in high-risk postmenopausal breast-cancer patients given adjuvant tamoxifen: Danish Breast Cancer Cooperative Group DBCG 82c randomised trial. Lancet. 1999 May 15;353(9165):1641-8. doi: 10.1016/S0140-6736(98)09201-0. PMID 10335782
- [Background] Ragaz J, Jackson SM, Le N, Plenderleith IH, Spinelli JJ, Basco VE, Wilson KS, Knowling MA, Coppin CM, Paradis M, Coldman AJ, Olivotto IA. Adjuvant radiotherapy and chemotherapy in node-positive premenopausal women with breast cancer. N Engl J Med. 1997 Oct 2;337(14):956-62. doi: 10.1056/NEJM199710023371402. PMID 9309100
- [Background] Heuts EM, van der Ent FW, von Meyenfeldt MF, Voogd AC. Internal mammary lymph drainage and sentinel node biopsy in breast cancer - A study on 1008 patients. Eur J Surg Oncol. 2009 Mar;35(3):252-7. doi: 10.1016/j.ejso.2008.06.1493. Epub 2008 Aug 5. PMID 18684584
- [Background] Farrus B, Vidal-Sicart S, Velasco M, Zanon G, Fernandez PL, Munoz M, Santamaria G, Albanell J, Biete A. Incidence of internal mammary node metastases after a sentinel lymph node technique in breast cancer and its implication in the radiotherapy plan. Int J Radiat Oncol Biol Phys. 2004 Nov 1;60(3):715-21. doi: 10.1016/j.ijrobp.2004.04.021. PMID 15465187
- [Background] TURNER-WARWICK RT. The lymphatics of the breast. Br J Surg. 1959 May;46:574-82. doi: 10.1002/bjs.18004620004. No abstract available. PMID 13839973
- [Background] Avisar E, Molina MA, Scarlata M, Moffat FL. Internal mammary sentinel node biopsy for breast cancer. Am J Surg. 2008 Oct;196(4):490-4. doi: 10.1016/j.amjsurg.2008.06.003. Epub 2008 Aug 23. PMID 18723148
- [Background] Veronesi U, Arnone P, Veronesi P, Galimberti V, Luini A, Rotmensz N, Botteri E, Ivaldi GB, Leonardi MC, Viale G, Sagona A, Paganelli G, Panzeri R, Orecchia R. The value of radiotherapy on metastatic internal mammary nodes in breast cancer. Results on a large series. Ann Oncol. 2008 Sep;19(9):1553-60. doi: 10.1093/annonc/mdn183. Epub 2008 May 7. PMID 18467318
- [Background] Freedman GM, Fowble BL, Nicolaou N, Sigurdson ER, Torosian MH, Boraas MC, Hoffman JP. Should internal mammary lymph nodes in breast cancer be a target for the radiation oncologist? Int J Radiat Oncol Biol Phys. 2000 Mar 1;46(4):805-14. doi: 10.1016/s0360-3016(99)00481-2. PMID 10705000
- [Background] Veronesi U, Marubini E, Mariani L, Valagussa P, Zucali R. The dissection of internal mammary nodes does not improve the survival of breast cancer patients. 30-year results of a randomised trial. Eur J Cancer. 1999 Sep;35(9):1320-5. doi: 10.1016/s0959-8049(99)00133-1. PMID 10658521
- [Background] Arriagada R, Le MG, Mouriesse H, Fontaine F, Dewar J, Rochard F, Spielmann M, Lacour J, Tubiana M, Sarrazin D. Long-term effect of internal mammary chain treatment. Results of a multivariate analysis of 1195 patients with operable breast cancer and positive axillary nodes. Radiother Oncol. 1988 Mar;11(3):213-22. doi: 10.1016/0167-8140(88)90003-5. PMID 3363169
- [Background] Cuzick J, Stewart H, Rutqvist L, Houghton J, Edwards R, Redmond C, Peto R, Baum M, Fisher B, Host H, et al. Cause-specific mortality in long-term survivors of breast cancer who participated in trials of radiotherapy. J Clin Oncol. 1994 Mar;12(3):447-53. doi: 10.1200/JCO.1994.12.3.447. PMID 8120544
- [Background] Hojris I, Overgaard M, Christensen JJ, Overgaard J. Morbidity and mortality of ischaemic heart disease in high-risk breast-cancer patients after adjuvant postmastectomy systemic treatment with or without radiotherapy: analysis of DBCG 82b and 82c randomised trials. Radiotherapy Committee of the Danish Breast Cancer Cooperative Group. Lancet. 1999 Oct 23;354(9188):1425-30. doi: 10.1016/s0140-6736(99)02245-x. PMID 10543669
- [Background] Darby SC, McGale P, Taylor CW, Peto R. Long-term mortality from heart disease and lung cancer after radiotherapy for early breast cancer: prospective cohort study of about 300,000 women in US SEER cancer registries. Lancet Oncol. 2005 Aug;6(8):557-65. doi: 10.1016/S1470-2045(05)70251-5. PMID 16054566
- [Background] Marks LB, Munley MT, Bentel GC, Zhou SM, Hollis D, Scarfone C, Sibley GS, Kong FM, Jirtle R, Jaszczak R, Coleman RE, Tapson V, Anscher M. Physical and biological predictors of changes in whole-lung function following thoracic irradiation. Int J Radiat Oncol Biol Phys. 1997 Oct 1;39(3):563-70. doi: 10.1016/s0360-3016(97)00343-x. PMID 9336133
- [Background] Kahan Z, Csenki M, Varga Z, Szil E, Cserhati A, Balogh A, Gyulai Z, Mandi Y, Boda K, Thurzo L. The risk of early and late lung sequelae after conformal radiotherapy in breast cancer patients. Int J Radiat Oncol Biol Phys. 2007 Jul 1;68(3):673-81. doi: 10.1016/j.ijrobp.2006.12.016. Epub 2007 Mar 9. PMID 17350177
- [Background] Kwa SL, Lebesque JV, Theuws JC, Marks LB, Munley MT, Bentel G, Oetzel D, Spahn U, Graham MV, Drzymala RE, Purdy JA, Lichter AS, Martel MK, Ten Haken RK. Radiation pneumonitis as a function of mean lung dose: an analysis of pooled data of 540 patients. Int J Radiat Oncol Biol Phys. 1998 Aug 1;42(1):1-9. doi: 10.1016/s0360-3016(98)00196-5. PMID 9747813
- [Background] Lind PA, Marks LB, Hardenbergh PH, Clough R, Fan M, Hollis D, Hernando ML, Lucas D, Piepgrass A, Prosnitz LR. Technical factors associated with radiation pneumonitis after local +/- regional radiation therapy for breast cancer. Int J Radiat Oncol Biol Phys. 2002 Jan 1;52(1):137-43. doi: 10.1016/s0360-3016(01)01715-1. PMID 11777631
- [Background] Wennberg B, Gagliardi G, Sundbom L, Svane G, Lind P. Early response of lung in breast cancer irradiation: radiologic density changes measured by CT and symptomatic radiation pneumonitis. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1196-206. doi: 10.1016/s0360-3016(01)02770-5. PMID 11955730
- [Background] N. Xu, M. Ho, C.G. Morris, N.P. Mendenhall. Proton treatment of peripheral lymph nodes in breast cancer. Int J Radiat Oncol Biol Phys 2010; 78: S803.
- See also: University of Florida Proton Therapy Institute website — http://www.floridaproton.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Phase: During this phase, each patient will have both a proton and conventional radiation plan performed. The superior plan in regard to minimizing dose to heart will be the plan actually chosen for treating the patient.
- Conventional Photon Plan: Conventional (photon): 50.4 Gray (Gy) to the breast/chest wall and peripheral lymph nodes at 1.8 Gy per fraction
  This number will automatically be equal to 0 during the 'induction phase' period and will only have a count in the 'treatment phase' period if a patient was actually assigned to this treatment.
- 3D-Proton/Conventional Plan or 3D-proton Only: 3D-Proton/Conventional plan or 3D-proton only: 50.4 Cobalt Gray Equivalent (CGE)/Gray (Gy) to the breast/chest wall and peripheral lymph nodes at 1.8 CGE/Gy
  This number will automatically be equal to 0 during the 'induction phase' period and will only have a count in the 'treatment phase' period if a patient was actually assigned to this treatment.
Period: Induction Phase
Arm/Group | Induction Phase | Conventional Photon Plan | 3D-Proton/Conventional Plan or 3D-proton Only
Started | 18 | 0 | 0
Completed | 18 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Phase
Arm/Group | Induction Phase | Conventional Photon Plan | 3D-Proton/Conventional Plan or 3D-proton Only
Started | 0 | 0 | 18
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Breast Patients Planned With Both Proton & Conventional Plans: Each patient is planned with both proton and conventional plans and the superior plan is chosen for treatment.
  Conventional plan: 50.4 Gy to the breast/chest wall and peripheral lymph nodes at 1.8 Gy per fraction
  Proton plan: 50.4 Cobalt Gray Equivalent/Gray to the breast/chest wall and peripheral lymph nodes at 1.8 Cobalt Gray Equivalent/Gray per fraction
Arm/Group | Breast Patients Planned With Both Proton & Conventional Plans
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: Years] | 52 [37 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Volume of Heart Receiving ≥ 5 Gray (Gy)/Cobalt Gray Equivalent (CGE)
Description: A reduction of 50% in heart volume exposed to radiation doses ≥ 5 Gy/CGE was considered preferred outcome in this study plan.
Time Frame: 2 weeks prior to starting radiation therapy.
Measure: Median (Full Range); unit: % of heart receiving >= 5 Gray (Gy)
Groups:
- Conventional Photon Plan: Photon: 50.4 Gray (Gy) to the breast/chest wall and peripheral lymph nodes at 1.8 Gy per fraction
- 3D-Proton/Conventional Plan or 3D-proton Only: 3D-Proton/Conventional plan or 3D-proton only: 50.4 Cobalt Gray Equivalent (CGE)/Gray (Gy) to the breast/chest wall and peripheral lymph nodes at 1.8 CGE/Gy per fraction
Arm/Group | Conventional Photon Plan | 3D-Proton/Conventional Plan or 3D-proton Only
Number analyzed (Participants) | 18 | 18
% of heart receiving >= 5 Gray (Gy) | 34.7 [6.9 to 60.0] | 2.7 [0.1 to 12.3]
Statistical Analysis 1: Comparison: Conventional Photon Plan vs 3D-Proton/Conventional Plan or 3D-proton Only; Test type: Superiority or Other; p = 0.0078, Wilcoxon (Mann-Whitney); Non-parametric paired t-test (Wilcoxon) = 29.1

2. Secondary Outcome: Secondary Dosimetric Endpoint
Description: Assess improvements in other dosimetry endpoints including lung dose (mean lung dose, V20, V5), heart dose (mean heart, V20, V5), mean dose to the thyroid, mean esophageal dose, D95 coverage for axillary, supraclavicular and internal mammary nodes, maximal spinal cord dose (Dmax) and skin Dmax.
Time Frame: 2 weeks prior to starting radiation therapy.
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of Acute Side Effects
Description: Assess acute toxicities including pericarditis, pneumonitis, dermatitis, fatigue, and nausea.
Time Frame: Participants will be assessed weekly during radiation therapy for an expected average of 7 weeks.
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of Longterm Side Effects and Disease Specific End Points.
Description: Assess late toxicities including clinical and sub-clinical heart disease, pulmonary fibrosis, soft tissue fibrosis, rib fracture, and secondary malignancies.
  Analyze local control, progression-free survival, and overall survival.
Time Frame: 1 month following completion of treatment, then every 6 months for 5 years, then annually thereafter.
Reporting Status: Not Posted

5. Secondary Outcome: Assessment of Cardiac Function Markers
Description: Assess levels of cardiac function markers Troponin and Brain Naturietic Peptide before and after treatment.
Time Frame: after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From start of radiation therapy to date of last follow-up.
Groups:
- Breast Patients Planned With Both Proton & Conventional Plans: All patients ultimately treated under the proton plan, so the denominator for all adverse events refers exclusively to the proton arm and not conventional.
  Each patient was planned with both proton and conventional plans and the superior plan was chosen for treatment.
  Conventional plan: 50.4 Gy to the breast/chest wall and peripheral lymph nodes at 1.8 Gy per fraction
  Proton plan: 50.4 Cobalt Gray Equivalent/Gray to the breast/chest wall and peripheral lymph nodes at 1.8 Cobalt Gray Equivalent/Gray per fraction
Arm/Group | Breast Patients Planned With Both Proton & Conventional Plans
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Patients Planned With Both Proton & Conventional Plans (N=18)
Skin infection (Infections and infestations) | 2 (2) — All patients ultimately treated under the proton plan, so the denominator for this event refers exclusively to the proton arm and not conventional.
Radiation dermatitis (Injury, poisoning and procedural complications) | 4 (4) — All patients ultimately treated under the proton plan, so the denominator for this event refers exclusively to the proton arm and not conventional.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breast Patients Planned With Both Proton & Conventional Plans (N=18)
Breast atrophy (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 7 (7)
Wound infection (Infections and infestations) | 2 (2)
Lymphedema (Reproductive system and breast disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No